CLINICAL TRIAL: NCT01331577
Title: Psychoneuroendocrinological Efficacy Study of an Integrative-kinesiological to a Cognitive-behavioural Intervention With Healthy Individuals
Brief Title: Comparison of the Efficacy of an Integrative-kinesiological to a Cognitive-behavioural Intervention
Acronym: IKSIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IKSIT_2011
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Healthy; Primary Prevention; Stress; Kinesiology; cognitive behavioural therapy; Prevention

ARMS (3):
- Cognitive behavioural Intervention (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Training
- Integrative Kinesiology Intervention (Experimental)
  Interventions: Behavioral: Integrative Kinesiology Intervention
- Waiting-List control group (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Training — Two day seminar
  Arms: Cognitive behavioural Intervention
Behavioral: Integrative Kinesiology Intervention — Two day seminar
  Arms: Integrative Kinesiology Intervention

SUMMARY:
Stress is a common problem with significant consequences for health. It can be a trigger for somatic diseases as well as psychological disorders and leads through missed working days and healthcare cost to a high economic loss. It is for health and economic reasons essential to develop and evaluate effective interventions that can inoculate against stress and build inner strength.

A cognitive-behavioural training for groups that is well evaluated and has shown to be effective is the Stress-Inoculation-Training by Meichenbaum. As the public utilization of methods of the complementary and alternative medicine is increasing a rigorous evaluation is needed. Integrative Kinesiology is a popular method that has been said to be effective against stress and its symptoms.

The investigators propose a randomized controlled evaluation and comparison of the interventions to each other and to a waiting-list control group. Hypothesis: Healthy volunteers attending a two dayseminar will show significantly reduced psychobiological reactivity, decreased stress perception and less anxiety to a standardized psychosocial stress test compared to the waiting list group. A total of 64 healthy volunteers will be randomly assigned to one of the three groups. The efficacy of the interventions will be measured through the Trier Social Stress Test (TSST) to measure the psychobiological stress reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Ready to participate in randomly one of the three groups
* mentally and physically healthy
* Sufficient German-speaking abilities to participate in the training

Exclusion Criteria:

* previous experience with Integrative Kinesiology or cognitive-behavioural therapy
* previous experience with the Trier Social Stress Test
* daily alcohol consumption: > two alcoholic drinks
* daily tobacco consumption: > 5 cigarettes per day
* any kind of drug abuse
* pregnancy, after the second trimenon
* intake ofe hormonal compounds (birth control pill and hormon replacement therapy)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area under curve with respect to increase of salivary cortisol titer | 8x during TSST
  TSST evaluation day will take place between 2 weeks and one month on average after the treatments are finished.
  Trier Social Stress Tests procedure will last close to two hours. Samples are collected at: T + 02; +25; +38; +48; +58; + 1:08; +1:23; + 1.38

SECONDARY OUTCOMES:
Salivary alpha amylase reactivity to the TSST | 8x during TSST
  TSST evaluation day will take place between 2 weeks and one month on average after the treatments are finished.
  Trier Social Stress Tests procedure will last close to two hours. Samples are collected at: T + 02; +25; +38; +48; +58; + 1:08; +1:23; + 1.38
Sense of Coherence | Baseline, post intervention and follow up
  Baseline: After recruitment and acceptance to the study Post: One week after the training is fulfilled Follow-up: One week after the TSST
  Measured by: Sense of Coherence questionnaire (SOC-L9)
Perceived Stress | Baseline, post intervention and follow up
  Baseline: After recruitment and acceptance to the study Post: One week after the training is fulfilled Follow-up: One week after the TSST
  Measured by: Perceived Stress Scale (PSS)
self efficacy expectancy | Baseline, post intervention and follow up
  Baseline: After recruitment and acceptance to the study Post: One week after the training is fulfilled Follow-up: One week after the TSST
  Measured by: Self-efficacy-expectancy questionnaire (SWE)

CONTACTS AND LOCATIONS:
Overall Officials: Lars B. Sonderegger, Principal Investigator — University of Zurich; Reinhard Saller, Prof., Study Chair — University of Zurich; Ulrike Ehlert, Prof., Study Chair — University of Zurich
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland